CLINICAL TRIAL: NCT01482273
Title: The BERN Ultrasound-enhanced Thrombolysis for Ilio-Femoral Deep Vein Thrombosis versUs Standard Catheter Directed thromboLysis Trial (BERNUTIFUL-Trial)
Brief Title: Ultrasound-enhanced Thrombolysis Versus Standard Catheter Directed Thrombolysis for Ilio-femoral Deep Vein Thrombosis
Acronym: BERNUTIFUL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Nils Kucher, Division of Clinical and Interventional Angiology, Swiss Cardiovascular Center, University Hospital and University of Bern
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150/11
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Venous Thrombosis; Postthrombotic Syndrome
Keywords: catheter-directed thrombolysis; ilio-femoral deep vein thrombosis; Postthrombotic syndrome; Phlebographic scores; Phlebography; Catheters
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDT+US group (Active Comparator): CDT using the EkoSonic Endovascular System with intravascular high-frequency, low-power ultrasound for 15 hours.
  Interventions: Procedure: CDT+US group
- CDT-US group (Active Comparator): CDT using the EkoSonic Endovascular System without intravascular high-frequency, low-power ultrasound for 15 hours.
  Interventions: Procedure: CDT-US group

INTERVENTIONS:
Procedure: CDT+US group — CDT using the EkoSonic Endovascular System with intravascular high-frequency, low-power ultrasound for 15 hours.
  Arms: CDT+US group
Procedure: CDT-US group — CDT using the EkoSonic Endovascular System without intravascular high-frequency, low-power ultrasound for 15 hours.
  Arms: CDT-US group

SUMMARY:
Patients with deep vein thrombosis (DVT) of the ilio-femoral veins have increased risk for developing post-thrombotic syndrome (PTS) and recurrent venous thromboembolism compared to more distal DVT. There's evidence that the early removal of the obstructing thrombus by catheter directed thrombolysis (CDT) reduces the risk of developing a PTS, and a higher degree of thrombolysis is associated with lower incidence of PTS, better quality of life and lower risk of recurrent venous thromboembolism. A further development is ultrasound-enhanced thrombolysis combining CDT with a sophisticated catheter system that employs high-frequency, low-dose ultrasound. In vitro experiments showed that adding ultrasound to thrombolytic drugs accelerates thrombolysis while Ultrasound exposure alone results in no thrombolysis, however the superiority of ultrasound-enhanced thrombolysis over standard CDT has never been formally assessed in vivo. The hypothesis for this study is that ultrasound-enhanced thrombolysis reaches a higher degree of thrombolysis than standard CDT in patients with symptomatic ilio-femoral DVT.

DETAILED DESCRIPTION:
Background

Deep vein thrombosis (DVT) is a public health problem with an annual incidence of 1 per 1000. Besides the acute risk of potentially fatal pulmonary embolism or phlegmasia cerulea dolens, these patients are at increased risk of recurrent venous thromboembolism, and in the long term 20-40% of them develop a post-thrombotic syndrome (PTS). PTS mainly develops in patients with DVT affecting the ilio-femoral veins, adversely affects the quality of life and causes important health care costs to the society. There's evidence that the early removal of the obstructing thrombus reduces the risk of developing a PTS, and a higher degree of thrombolysis is associated with lower incidence of PTS, better quality of life and lower risk of recurrent venous thromboembolism. Therefore, in addition to standard anticoagulation therapy, the latest international guidelines recommend catheter-directed thrombolysis (CDT) as first-line treatment for patients with ilio-femoral DVT and low bleeding risk. CDT refers to the infusion of thrombolytic drugs directly into the thrombus via a multisidehole catheter which is embedded in the thrombus using imaging guidance. A further development is ultrasound-enhanced thrombolysis combining CDT with a sophisticated catheter system that employs high-frequency, low-dose ultrasound. In vitro experiments showed that adding Ultrasound to thrombolytic drugs accelerates thrombolysis while Ultrasound exposure alone results in no thrombolysis. Although ultrasound-enhanced thrombolysis is now widely used to treat ilio-femoral DVT or high-risk pulmonary embolism, it is currently not known if this technique is superior to standard CDT.

Objective

To determine if the addition of intravascular high-frequency/low-dose ultrasound to standard CDT increases the percentage of clot lysis compared to CDT alone after treatment duration of 15 hours in patients with symptomatic ilio-femoral DVT and low bleeding risk

Methods

Study design: open-label (with blinding of data-analyzing physicians), randomized, controlled, single center clinical trial with a follow-up period of 12 months.

Subjects: total of 20 patients (10 in each study group) of 18-75 years of age with acute, symptomatic, objectively confirmed ilio-femoral DVT and a low bleeding risk.

Intervention: CDT using the EkoSonic Endovascular System with (CDT+US group) or without (CDT-US group) intravascular high-frequency, low-power ultrasound for 15 hours.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic proximal DVT involving the iliac and/or common femoral vein, confirmed by Duplex Sonography, Angio-CT, Angio-MRI or Phlebography
* Written informed consent

Exclusion Criteria

* Age less than 18 years or greater than 75 years
* Symptom duration > 14 days for the DVT episode in the index leg (i.e., non-acute DVT).
* In the index leg: established post-thrombotic syndrome (PTS) or previous symptomatic DVT within the last 2 years.
* Limb-threatening circulatory compromise.
* PE with hemodynamic compromise (i.e., hypotension).
* Inability to tolerate catheter procedure due to severe dyspnea or acute systemic illness.
* Allergy, hypersensitivity, or thrombocytopenia from heparin, r-tPA, or iodinated contrast, except for mild-moderate contrast allergies for which steroid pre-medication can be used.
* Known significant bleeding risk, or known coagulation disorder (including vitamin K antagonists with INR > 2.0 and platelet count < 100 000/mm3)
* Severe renal impairment (estimated GFR < 30 ml/min).
* Active bleeding, recent (< 3 mo) GI bleeding, severe liver dysfunction, bleeding diathesis.
* Recent (< 3 mo) internal eye surgery or hemorrhagic retinopathy; recent (< 10 days) major surgery, cataract surgery, trauma, CPR, obstetrical delivery, or other invasive procedure.
* History of stroke or intracranial/intraspinal bleed, tumor, vascular malformation, aneurysm.
* Severe hypertension on repeated readings (systolic > 180 mmHg or diastolic > 105 mmHg).
* Pregnant, lactation or parturition within the previous 30 days (positive pregnancy test, women of childbearing age must be tested or use a medically accepted method of birth control).
* Recently (< 1 mo) had thrombolysis.
* Life expectancy < 6 months or chronic non-ambulatory status.
* Participating in any other investigational drug or device study or previous enrollment in this study
* Inability to provide informed consent or to comply with study assessments (e.g. due to cognitive impairment or geographic distance).
* Any other condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Improvement of Total EKOS Thrombus Score, a specifically developed venographic scoring system | After 15 hours of CDT

SECONDARY OUTCOMES:
Improvement of the "Venous Registry Index" venographic scoring system | After 15 hours of CDT
Early symptom relief assessed by standardized limb circumference measurements and validated visual analogue pain scale | During and after 15 hours of CDT
Treatment related complications | 30 days
Development of PTS assessed by Villalta scale and Quality of life (CIVIQ) | After 12 months
Venous valve patency/insufficiency assessed by duplex sonography | After 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nils Kucher, MD, Principal Investigator — Division of Clinical and Interventional Angiology, Swiss Cardiovascular Center, University Hospital and University of Bern; Torsten Willenberg, MD, Study Director — Division of Clinical and Interventional Angiology, Swiss Cardiovascular Center, University Hospital and University of Bern; Iris Baumgartner, MD, Study Director — Division of Clinical and Interventional Angiology, Swiss Cardiovascular Center, University Hospital and University of Bern; Rolf P Engelberger, MD, Study Director — Division of Clinical and Interventional Angiology, Swiss Cardiovascular Center, University Hospital and University of Bern
Locations (1):
- Division of Clinical and Interventional Angiology, Swiss Cardiovascular Center, University Hospital and University of Bern, Bern, Switzerland

REFERENCES:
- [Background] Jaff MR, McMurtry MS, Archer SL, Cushman M, Goldenberg N, Goldhaber SZ, Jenkins JS, Kline JA, Michaels AD, Thistlethwaite P, Vedantham S, White RJ, Zierler BK; American Heart Association Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; American Heart Association Council on Peripheral Vascular Disease; American Heart Association Council on Arteriosclerosis, Thrombosis and Vascular Biology. Management of massive and submassive pulmonary embolism, iliofemoral deep vein thrombosis, and chronic thromboembolic pulmonary hypertension: a scientific statement from the American Heart Association. Circulation. 2011 Apr 26;123(16):1788-830. doi: 10.1161/CIR.0b013e318214914f. Epub 2011 Mar 21. PMID 21422387
- [Background] Siddiqi F, Odrljin TM, Fay PJ, Cox C, Francis CW. Binding of tissue-plasminogen activator to fibrin: effect of ultrasound. Blood. 1998 Mar 15;91(6):2019-25. PMID 9490686
- [Background] Engelhardt TC, Taylor AJ, Simprini LA, Kucher N. Catheter-directed ultrasound-accelerated thrombolysis for the treatment of acute pulmonary embolism. Thromb Res. 2011 Aug;128(2):149-54. doi: 10.1016/j.thromres.2011.05.014. Epub 2011 Jun 8. PMID 21641020
- [Result] Kahn SR, Shrier I, Julian JA, Ducruet T, Arsenault L, Miron MJ, Roussin A, Desmarais S, Joyal F, Kassis J, Solymoss S, Desjardins L, Lamping DL, Johri M, Ginsberg JS. Determinants and time course of the postthrombotic syndrome after acute deep venous thrombosis. Ann Intern Med. 2008 Nov 18;149(10):698-707. doi: 10.7326/0003-4819-149-10-200811180-00004. PMID 19017588
- [Result] Popuri RK, Vedantham S. The role of thrombolysis in the clinical management of deep vein thrombosis. Arterioscler Thromb Vasc Biol. 2011 Mar;31(3):479-84. doi: 10.1161/ATVBAHA.110.213413. PMID 21325669
- [Result] Grewal NK, Martinez JT, Andrews L, Comerota AJ. Quantity of clot lysed after catheter-directed thrombolysis for iliofemoral deep venous thrombosis correlates with postthrombotic morbidity. J Vasc Surg. 2010 May;51(5):1209-14. doi: 10.1016/j.jvs.2009.12.021. Epub 2010 Mar 27. PMID 20347543
- [Result] Grommes J, Strijkers R, Greiner A, Mahnken AH, Wittens CH. Safety and feasibility of ultrasound-accelerated catheter-directed thrombolysis in deep vein thrombosis. Eur J Vasc Endovasc Surg. 2011 Apr;41(4):526-32. doi: 10.1016/j.ejvs.2010.11.035. Epub 2011 Jan 21. PMID 21256773
- [Result] Hull RD, Marder VJ, Mah AF, Biel RK, Brant RF. Quantitative assessment of thrombus burden predicts the outcome of treatment for venous thrombosis: a systematic review. Am J Med. 2005 May;118(5):456-64. doi: 10.1016/j.amjmed.2005.01.025. PMID 15866245
- [Result] Sharifi M, Mehdipour M, Bay C, Smith G, Sharifi J. Endovenous therapy for deep venous thrombosis: the TORPEDO trial. Catheter Cardiovasc Interv. 2010 Sep 1;76(3):316-25. doi: 10.1002/ccd.22638. PMID 20578224
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829
- [Derived] Broderick C, Watson L, Armon MP. Thrombolytic strategies versus standard anticoagulation for acute deep vein thrombosis of the lower limb. Cochrane Database Syst Rev. 2021 Jan 19;1(1):CD002783. doi: 10.1002/14651858.CD002783.pub5. PMID 33464575
- [Derived] Engelberger RP, Stuck A, Spirk D, Willenberg T, Haine A, Periard D, Baumgartner I, Kucher N. Ultrasound-assisted versus conventional catheter-directed thrombolysis for acute iliofemoral deep vein thrombosis: 1-year follow-up data of a randomized-controlled trial. J Thromb Haemost. 2017 Jul;15(7):1351-1360. doi: 10.1111/jth.13709. Epub 2017 Jun 5. PMID 28440041
- [Derived] Engelberger RP, Spirk D, Willenberg T, Alatri A, Do DD, Baumgartner I, Kucher N. Ultrasound-assisted versus conventional catheter-directed thrombolysis for acute iliofemoral deep vein thrombosis. Circ Cardiovasc Interv. 2015 Jan;8(1):e002027. doi: 10.1161/CIRCINTERVENTIONS.114.002027. PMID 25593121